CLINICAL TRIAL: NCT04433962
Title: Investigation of the Effects of Balance Training on Balance and Functional Status Patients With Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nuray Elibol, Assistant of Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/22-01
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Arthroplasty Complications; Physical Disability; Osteoarthritis, Hip
Keywords: osteoarthritis; hip; total hip arthroplasty; balance training; function; assessment
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional rehabilitation group (Active Comparator): the conventional rehabilitation group completed hip joint range of motion and muscle strengthening exercises
  Interventions: Other: Exercise training
- conventional rehabilitation + balance training group (Experimental): The conventional rehabilitation + balance training group completed hip joint range of motion and muscle strengthening exercises and 12 balance exercises.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training
  Other Names: conventional rehabilitation; conventional rehabilitation and balance training

SUMMARY:
The purpose of this study is to investigate the effects of balance training in patients with THA until 26 weeks postoperatively. Thirty-two patients with hip osteoarthritis who were candidates for THA were recruited to the study. Sixteen patients with THA completed the study protocol and the patients were randomized into 2 groups: conventional rehabilitation (CR, n=8) or conventional rehabilitation plus balance training (CR + BT, n=8) groups. The patients were evaluated by hand-held dynamometer, single leg stance test (SLST), Tetrax balance system, Harris hip score, lower extremity function scale, 5 times sit-to-stand test and 50 foot timed walk test preoperatively and in the 8th, 14th and 26th weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty due to osteoarthritis
* First time hip surgery/prothesis
* no involvement in any exercise program in the past 12 months

Exclusion Criteria:

* THA due to hip fracture,
* revision hip prothesis,
* arthritis in other joints limited function
* neurologic problems that limited function and balance,
* body mass index greater than 40 kg/m2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2016-12-25 (Actual)

PRIMARY OUTCOMES:
single leg test | Pre-op to post-op 26. week
  Patients were tested first with eyes opened and then with eyes closed; they were asked to stand on either their left or right leg and tried to keep their legs from touching and to maintain single-leg stance for as long as possible. The test and time began once the foot was lifted off the floor, and ended when placing the lifted foot on the floor or with arm movements. The test was terminated following a maximum of 45 s, and each leg was tested three times with eyes opened and eyes closed and the best of the three trials were recorded
Tetrax Balance Assessment | Pre-op to post-op 26. week
  Tetrax Balance Assessment System (Sunlight Medical Ltd.Ramat Gan, Israel); is a valid, reliable and objective method to evaluate balance and fall risk. The system obtains data by using 4 different platforms which measure vertical pressure fluctuations arising from two heels and two fingertips. Patients were instructed an immobile posture for 32 s for each of the eight sensory conditions.The fall risks of the patients were calculated as percentage (%) by a posturographic program considering the oscillation rates. A value between 0% and 36% is judged as mild risk; a value between 37% and 58%, as moderate risk; and between 59% and 100%, as high risk. The higher score is showed the greater falling risk
Sit to stand test | Pre-op to post-op 26. week
  STS; is an objective functional measure of strength correlating with ambulatory independence. Sit-to-stand (such as the 5 STS) activities are recommended as the minimal core set of performance-based outcome measures in OA research and clinical practice [21]. Patients sit on a height adjustable chair such that a 90⁰ angle is formed when the femur is horizontal and tibia vertical with their feet shoulder width apart and their arms crossed against their chest. Patients are timed as they 5 times stand up from chair and sit down again without using their hand, time was recorded as second
50 feet walk test | Pre-op to post-op 26. week
  50 FWT; is a reliable measurement method and commonly used in studies of exercise based OA. All patients are asked to walk as quickly as possible in 50 feet length distance. The physiotherapist counted number of steps and as soon as the patient finished to walking 50 feet length distance and the time was recorded as seconds
Harris hip score | Pre-op to post-op 26. week
  Many different hip scoring scales are used in assessment of THA's results [23]. HHS is a joint specific outcome measurements and the most frequently used in assessment of THA patients. It has been used in a number of studies over the years and has been shown to have high validity and reliability [23,24]. HHS was recorded, a score commonly used in this context, which contains questions about pain, function, absence of deformity, and range-of-motion. The best possible score is 100 points
Lower extremity function scale | Pre-op to post-op 26. week
  is a region specific measure, was conceived to assess the lower extremity functional status of patients and the reliability estimates have been high when investigated in the THA and TKA population. The LEFS is composed of 20 items each scored on a 5 point adjectival scale with '0' extreme difficulty or unable to perform the activity and '4' no difficulty. The items are summed to produce a total LEFS score, which can vary from 0 to 80.

SECONDARY OUTCOMES:
Pain assessment | Pre-op to post-op 26. week
  Visual analog scale was used to determine to degree of pain. The patient was asked to choose a number 0 and 10 on a chart. 0 indicates "no pain" and 10 indicates "very severe pain".
Range of motion | Pre-op to post-op 26. week
  Hip extension, hipflexion, hip abduction and hip adduction was measured with goniometer.
Muscle strength | Pre-op to post-op 26. week
  Maximal isometric muscle strength was measured with a handheld dynamometer (HHD) (Lafayette Instrument Company).

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Elibol, PhD, Principal Investigator — Ege University
Locations (1):
- Dokuz Eylul University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No